CLINICAL TRIAL: NCT01232855
Title: Regulation of S100A10 by the PML-RAR-alpha Oncoprotein
Brief Title: Biomarkers in Tissue Samples From Patients With Acute Promyelocytic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML11B5; COG-AAML11B5 (Other: Children's Oncology Group); NCI-2011-02844 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML11B5 (Other: Children's Oncology Group)
Record Dates: First submitted 2010-10-30; First posted 2010-11-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute promyelocytic leukemia (M3); childhood acute promyelocytic leukemia (M3); adult acute myeloid leukemia in remission; untreated adult acute myeloid leukemia; childhood acute myeloid leukemia in remission; untreated childhood acute myeloid leukemia and other myeloid malignancies
MeSH Terms: conditions — Leukemia; Leukemia, Promyelocytic, Acute | interventions — Blotting, Western; Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: protein expression analysis
Genetic: western blotting
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples fo tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in tissue samples from patients with acute promyelocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Demonstrate that S100A10 is expressed on APL cells and that levels of S100A10 correspond to the amount of fibrinolytic activity.
* Evaluate the impact of ATRA on S100A10 level and fibrinolytic activity in vitro.
* Evaluate the impact of S100A10 knockdown on fibrinolytic activity.
* Correlate in vitro findings in cell culture to primary patient samples both pre- and post-ATRA therapy.

OUTLINE: This is a multicenter study.

Previously collected samples are analyzed via flow cytometry and western blot analysis. Cell surface levels of S100A10 and annexin A2 are correlated to the promyelocyte population and total protein levels are examined to determine total annexin A2 and S100A10 in acute promyelocytic leukemia cells.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute promyelocytic leukemia
* Available cryopreserved cells from diagnosis or cryopreserved cells from remission (germline)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients With Acute Promyelocytic Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Demonstration that S100A10 is expressed on acute promyelocytic leukemia cells and that levels of S100A10 correspond to the amount of fibrinolytic activity
Evaluation of the impact of all-trans retinoic acid (ATRA) on S100A10 level and fibrinolytic activity in vitro
Evaluation of the impact of S100A10 knockdown on fibrinolytic activity
Correlation of in vitro findings in cell culture to primary patient samples both pre- and post-ATRA therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jason N. Berman, MD, Principal Investigator — IWK Health Centre